CLINICAL TRIAL: NCT07045883
Title: Mechanism and Clinical Application of Vitamin D in Influencing the Prognosis of Idiopathic Sudden Sensorineural Hearing Loss
Brief Title: Mechanism and Application of Vitamin D in Idiopathic Sudden Sensorineural Hearing Loss
Acronym: N
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024QNB016; 2024QNB016 (Other Grant/Funding Number: Science and Education Division, Fujian Provincial Health Commission)
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Sudden Sensorineural Hearing Loss
Keywords: Idiopathic sudden sensorineural hearing loss; vitamin D; 25（OH）D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D Supplementation (Experimental): Participants receive Vitamin D3 (dose: 800 IU/day, orally, for 4 weeks)
  Interventions: Drug: Vitamin D Supplementation+ standard treatment
- Standard Care (Other): Standard treatment
  Interventions: Other: standard treatment

INTERVENTIONS:
Drug: Vitamin D Supplementation+ standard treatment — The experimental group was tested for 25(OH)D concentration after enrollment, and the experimental group was divided into vitamin D deficiency group and vitamin D normal group. In the vitamin D-deficient group, participants will receive standard treatment plus oral vitamin D3 supplementation (800 IU daily for 4 weeks), whereas the vitamin D normal group will receive standard treatment alone
  Arms: Vitamin D Supplementation
Other: standard treatment — The experimental group was tested for 25(OH)D concentration after enrollment, and the experimental group was divided into vitamin D deficiency group and vitamin D normal group. The vitamin D normal group will receive standard treatment alone
  Arms: Standard Care

SUMMARY:
Clinical Trial Protocol: Investigating the Therapeutic Efficacy of Vitamin D in ISSNHL。Core Research Questions Can vitamin D supplementation improve the prognosis of Idiopathic Sudden Sensorineural Hearing Loss (ISSNHL)? What potential medical issues might arise during vitamin D administration? Study Design

A controlled trial comparing:

Intervention group: Vitamin D supplementation + standard care Control group: Standard care alone Participant Procedures

Baseline assessment:

Venous blood draw (2 mL) for 25(OH)D level measurement. intervention phase:Daily vitamin D supplementation for 1 month

Endpoint evaluation (1-month follow-up):

Repeat audiometric testing (pure-tone audiometry). Post-treatment 25(OH)D concentration analysis.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Idiopathic Sudden Sensorineural Hearing Loss First-time unilateral occurrence Illness duration ≤14 days No prior treatment

Exclusion Criteria:

Middle ear lesions, inner ear malformations, or retrocochlear lesion Age <18 years, pregnant or lactating women History of ear surgery or familial hereditary deafness With osteoporosis, osteochondrosis, rickets and other systemic serious systemic diseases Those who refuse to be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin D deficiency as a prognostic factor in ISSNHL | From enrollment to the end of follow-upt at 14 weeks
  Plasma 25(OH)D concentrations of all enrolled cases in the experimental group and the healthy control group were compared to explore whether 25(OH)D differed in the idiopathic sudden deafness group and with the healthy control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital of Xiamen University, School of Medicine, Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No